CLINICAL TRIAL: NCT02089815
Title: Effectiveness of a Simple Designed Programme of Home Based Exercise in Preventing Fall and Improving Balance and Strength in Older People With Mild to Moderate Balance Dysfunction: A Randomized Controlled Trials
Brief Title: Home Based Exercise in Preventing Fall and Improving Balance in Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Chitima Boongird, Doctor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01-56-37
Record Dates: First submitted 2014-03-10; First posted 2014-03-18 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Patient Fall; Muscle Balance; Fear of Falling; Quality of Life
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Home based exercise (Experimental): simple designed home based exercise program
  Interventions: Behavioral: Home based exercise; Other: fall prevention education and counseling
- fall prevention education and counseling (Active Comparator): fall prevention education & counseling : home modification, vision screening, avoid sedative drugs use, proper shoes, report dizziness and fall to doctors
  Interventions: Other: fall prevention education and counseling

INTERVENTIONS:
Behavioral: Home based exercise — modified Otago exercise program to simple designed home based exercise program
  Other Names: combination strengthening and balance training program
  Arms: Home based exercise
Other: fall prevention education and counseling

SUMMARY:
Prior studies have shown multifaceted falls prevention program with home-based exercise reduced falls significantly in the community setting. The Otago exercise program has been tested in four separated controlled trials of community living people in New Zealand. Falls were the main outcome in each trail and were defined as "unintentionally coming to rest on the ground, floor or other lower level". Not only this combination strengthening and balance training exercise could reduce fall but also could benefit in cost-effectiveness for fall prevention and decrease mortality in those 80 and older. However the limitation of Otago exercise program is that the program was needed to be trained by skill nurses or physical therapists. There are 17 steps levels to adhere the program. As some studies have shown that fall prevention program adherence could be as low as 10-40%. In Thailand the lack of medical staffs are continued the problem in the community. Therefore to establish fall prevention guideline that will be suitable and translated into the real setting, this study is aimed to test the effectiveness of simple program home-based exercise comparing to non-simple program home based exercise in preventing fall and improve muscle strength and balance dysfunction in older people with mild to moderate balance dysfunction. The method is the randomized controlled trails.

ELIGIBILITY:
Inclusion Criteria:

1. Thai elderly aged 65 years or older
2. able to communicate and follow the home-based exercise programme
3. mild to moderate balance dysfunctions as followings:

   * functional reach test score less than 26 cm.
   * five time sit to stand test more than 17.9 seconds
   * able to walk independently or walk with only single cane
4. non diagnosed with moderate to severe dementia or depression
5. non diagnosed with parkinson disease
6. non diagnosed with cerebrovascular disease with less than grade 4 hemiparesis.
7. non diagnosed with acute arthritis or recent diagnosed within 6 months.
8. informed and consent to participate in the study
9. not participate in regular Tai-chi or Yoga exercise training.

Exclusion criteria:

1. Participants would like to withdraw from the study.
2. severe injury occured after following simple designed exercise program eg. tendon injuries.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 439 (Actual)
Dates: Start 2013-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
number of falls | 1 year
  Number of falls were measured at baseline, 12 weeks, 24 weeks and 1 year. At baseline, the participants will be interviewed the number of falls that occurred in the past 1 year period before enrollment.

SECONDARY OUTCOMES:
muscle strength | baseline, 12 weeks and 24 weeks
  There are two Measurements as following:
  1. Five time sit to stand test The participant stood up and sat down as quickly as possible from standard chair (47 cm high) 5 times, with arms folded across the chest.
  2. Timed up and go test The time required to rise from a chair, walk 3 meters distance, turn around, walk back and sit down.
Balance | Baseline, 12 weeks and 24 weeks
  The participants will be tested their balances by using Short form of Berg Balance scale (7 items, 0-28 scores.)

OTHER OUTCOMES:
fear of falling | baseline and at 24 weeks.
  Thai Falls efficacy scale-international (FES-I)
Quality of life | 1 year
  The participants will be interviewed by using Thai EQ-5D questionaires.

CONTACTS AND LOCATIONS:
Overall Officials: Chitima Boongird, MD, Principal Investigator — Department of Family Medicine, Ramathibodi Hospital, Mahidol University
Locations (1):
- Ramathibodi Hospital, Mahidol University, Bangkok, Bangkok, Thailand

REFERENCES:
- [Background] Day L. The Otago strength and balance exercise programme lowers the risk of death and falls in the older people at 12 months. Evid Based Nurs. 2011 Jul;14(3):76-8. doi: 10.1136/ebn1157. Epub 2011 Mar 24. No abstract available. PMID 21436159
- [Background] Kuptniratsaikul V, Praditsuwan R, Assantachai P, Ploypetch T, Udompunturak S, Pooliam J. Effectiveness of simple balancing training program in elderly patients with history of frequent falls. Clin Interv Aging. 2011;6:111-7. doi: 10.2147/CIA.S17851. Epub 2011 May 6. PMID 21594001
- [Background] Yang XJ, Hill K, Moore K, Williams S, Dowson L, Borschmann K, Simpson JA, Dharmage SC. Effectiveness of a targeted exercise intervention in reversing older people's mild balance dysfunction: a randomized controlled trial. Phys Ther. 2012 Jan;92(1):24-37. doi: 10.2522/ptj.20100289. Epub 2011 Oct 6. PMID 21979272
- [Background] Campbell AJ, Robertson MC, Gardner MM, Norton RN, Tilyard MW, Buchner DM. Randomised controlled trial of a general practice programme of home based exercise to prevent falls in elderly women. BMJ. 1997 Oct 25;315(7115):1065-9. doi: 10.1136/bmj.315.7115.1065. PMID 9366737
- [Background] Sherrington C, Whitney JC, Lord SR, Herbert RD, Cumming RG, Close JC. Effective exercise for the prevention of falls: a systematic review and meta-analysis. J Am Geriatr Soc. 2008 Dec;56(12):2234-43. doi: 10.1111/j.1532-5415.2008.02014.x. PMID 19093923
- [Background] Simek EM, McPhate L, Haines TP. Adherence to and efficacy of home exercise programs to prevent falls: a systematic review and meta-analysis of the impact of exercise program characteristics. Prev Med. 2012 Oct;55(4):262-275. doi: 10.1016/j.ypmed.2012.07.007. Epub 2012 Jul 17. PMID 22813920
- [Background] Howe TE, Rochester L, Neil F, Skelton DA, Ballinger C. Exercise for improving balance in older people. Cochrane Database Syst Rev. 2011 Nov 9;2011(11):CD004963. doi: 10.1002/14651858.CD004963.pub3. PMID 22071817
- [Background] Thomas S, Mackintosh S, Halbert J. Does the 'Otago exercise programme' reduce mortality and falls in older adults?: a systematic review and meta-analysis. Age Ageing. 2010 Nov;39(6):681-7. doi: 10.1093/ageing/afq102. Epub 2010 Sep 4. PMID 20817938
- [Background] Gates S, Fisher JD, Cooke MW, Carter YH, Lamb SE. Multifactorial assessment and targeted intervention for preventing falls and injuries among older people in community and emergency care settings: systematic review and meta-analysis. BMJ. 2008 Jan 19;336(7636):130-3. doi: 10.1136/bmj.39412.525243.BE. Epub 2007 Dec 18. PMID 18089892
- [Background] Gillespie LD, Robertson MC, Gillespie WJ, Lamb SE, Gates S, Cumming RG, Rowe BH. Interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD007146. doi: 10.1002/14651858.CD007146.pub2. PMID 19370674
- [Background] Day L, Fildes B, Gordon I, Fitzharris M, Flamer H, Lord S. Randomised factorial trial of falls prevention among older people living in their own homes. BMJ. 2002 Jul 20;325(7356):128. doi: 10.1136/bmj.325.7356.128. PMID 12130606
- [Background] Fabacher D, Josephson K, Pietruszka F, Linderborn K, Morley JE, Rubenstein LZ. An in-home preventive assessment program for independent older adults: a randomized controlled trial. J Am Geriatr Soc. 1994 Jun;42(6):630-8. doi: 10.1111/j.1532-5415.1994.tb06862.x. PMID 8201149
- [Background] Kimman M, Vathesatogkit P, Woodward M, Tai ES, Thumboo J, Yamwong S, Ratanachaiwong W, Wee HL, Sritara P. Validity of the Thai EQ-5D in an occupational population in Thailand. Qual Life Res. 2013 Aug;22(6):1499-506. doi: 10.1007/s11136-012-0251-2. Epub 2012 Aug 25. PMID 22926727
- [Background] Duncan PW, Weiner DK, Chandler J, Studenski S. Functional reach: a new clinical measure of balance. J Gerontol. 1990 Nov;45(6):M192-7. doi: 10.1093/geronj/45.6.m192. PMID 2229941
- [Background] Csuka M, McCarty DJ. Simple method for measurement of lower extremity muscle strength. Am J Med. 1985 Jan;78(1):77-81. doi: 10.1016/0002-9343(85)90465-6. PMID 3966492
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Chou CY, Chien CW, Hsueh IP, Sheu CF, Wang CH, Hsieh CL. Developing a short form of the Berg Balance Scale for people with stroke. Phys Ther. 2006 Feb;86(2):195-204. PMID 16445333
- [Background] Hill KD, Schwarz JA, Kalogeropoulos AJ, Gibson SJ. Fear of falling revisited. Arch Phys Med Rehabil. 1996 Oct;77(10):1025-9. doi: 10.1016/s0003-9993(96)90063-5. PMID 8857881